CLINICAL TRIAL: NCT01958476
Title: Improving Outcomes in Neonatal Abstinence Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA032889-01A1 (NIH)
Record Dates: First submitted 2013-08-14; First posted 2013-10-09 (Estimated); Results first posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-09

CONDITIONS: Neonatal Abstinence Syndrome; Neonatal Opioid Withdrawal
Keywords: Neonatal Abstinence Syndrome; Opioids
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Morphine; Methadone; Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neonatal Morphine Solution (Active Comparator): Infants randomized to this arm will receive neonatal morphine solution (0.2mg/mL) for first line therapy. Infants will be scored using the standardized Finnegan scoring system and will be initiated on treatment if they have 2 consecutive scores greater than or equal to 8 or 1 score greater than or equal to 12. Dosing will be weight and symptom based. A "double dummy" design will be used - each infant will be ordered for both a methadone/placebo study drug at 0.4 mg/mL and a morphine/placebo study drug at 0.2 mg/mL. Starting doses will range from 0.3mg/kg/day to 0.9mg/kg/day divided every 4 hours depending on the severity of the Finnegan scores. Doses will be increased to a maximum of 0.9mg/kg/day for continued scores generally >8 caused primarily by worsening NAS. Infants will be weaned by 10% of the maximum dose once every 24 - 48 hours and the medication will be discontinued once at 25% of the maximum dose.
  Interventions: Drug: Neonatal Morphine Solution; Drug: Phenobarbital
- Methadone (Active Comparator): Infants randomized to this group will receive methadone oral solution (0.4mg/mL) for first line therapy. Infants will be scored using the standardized Finnegan scoring system and will be initiated on treatment if they have 2 consecutive scores greater than or equal to 8 or 1 score greater than or equal to 12. Dosing will be weight and symptom based. Starting doses will range from 0.3mg/kg/day to 0.9mg/kg/day divided every 8 hours depending on the severity of the Finnegan scores. To maintain blinding of the two study arms, a "double dummy" design will be used - each infant will receive both methadone/placebo study drug at 0.4 mg/mL and a morphine/placebo study drug at 0.2 mg/mL. Doses will be increased to a maximum of 0.9mg/kg/day for continued scores generally >8 caused primarily by worsening NAS as needed. Infants will be weaned by 10% of the maximum dose once every 24-48 hours and the medication will be discontinued once at 25% of the maximum dose.
  Interventions: Drug: Methadone; Drug: Phenobarbital

INTERVENTIONS:
Drug: Neonatal Morphine Solution — Infants randomized to this arm will receive neonatal morphine solution (0.2mg/mL) for first line therapy. Infants will be scored using the standardized Finnegan scoring system and will be initiated on treatment if they have 2 consecutive scores greater than or equal to 8 or 1 score greater than 12. Dosing will be weight and symptom based. A "double dummy" design will be used - each infant will be ordered for both a methadone/placebo study drug at 0.4 mg/mL and a morphine/placebo study drug at 0.2 mg/mL. Starting doses will range from 0.3mg/kg/day to 0.9mg/kg/day divided every 4 hours depending on the severity of the Finnegan scores. Doses will be increased to a maximum of 0.9mg/kg/day for continued scores generally >8 caused primarily by worsening NAS. Infants will be weaned by 10% of the maximum dose once every 24 - 48 hours and the medication will be discontinued once at 25% of the maximum dose.
  Other Names: Morphine sulfate
  Arms: Neonatal Morphine Solution
Drug: Methadone — Infants randomized to this group will receive methadone oral solution (0.4mg/mL) for first line therapy. Infants will be scored using the standardized Finnegan scoring system and will be initiated on treatment if they have 2 consecutive scores greater than or equal to 8 or 1 score greater than or equal to 12. Dosing will be weight and symptom based. Starting doses will range from 0.3mg/kg/day to 0.9mg/kg/day divided every 8 hours depending on the severity of the Finnegan scores. To maintain blinding of the two study arms, a "double dummy" design will be used - each infant will receive both methadone/placebo study drug at 0.4 mg/mL and a morphine/placebo study drug at 0.2 mg/mL. Doses will be increased to a maximum of 0.9mg/kg/day for continued scores generally >8 caused primarily by worsening NAS as needed. Infants will be weaned by 10% of the maximum dose once every 24-48 hours and the medication will be discontinued once at 25% of the maximum dose.
  Other Names: Methadone oral solution
  Arms: Methadone
Drug: Phenobarbital — A second line medication will be added once the infant reaches maximum doses of the study drug (morphine or methadone) for continued scores generally >8. Infants will be loaded with 20mg/kg of phenobarbital with the option to re-load with 10mg/kg q8-12 hours for 2 more doses if needed for continued high scores. Maintenance therapy of 5mg/kg/day will be initiated 12 - 24 hours after the last loading dose. Phenobarbital trough levels will be monitored with goal levels of 20 - 30 mcg/mL.
  Phenobarbital will be weaned only after the infant has been weaned off of the study drug. Weaning will begin 48 hours after the study drug has been stopped by 20% of the maximum total daily dose every 3 days for scores <8. An infant may be discharged home 48 - 72 hours after the first wean. The remaining wean will be outlined in the discharge prescription, and followed up on by study staff with the goal of the phenobarbital discontinuation within a 2 week period.

SUMMARY:
1: SPECIFIC Aim I: To compare treatment options for neonatal abstinence syndrome (NAS) due to in-utero narcotic exposure. One hundred eighty four full-term infants with a diagnosis of NAS requiring medications will be studied. Infants will be randomized to receive either morphine or methadone. It is hypothesized that morphine treated infants will do better and require fewer days in the hospital compared to methadone treated infants.

2. SPECIFIC Aim II: To evaluate the effects of NAS treatment on long-term neurodevelopmental outcome. Infants will be evaluated with development testing at 18 months of age. It is hypothesized that morphine treated infants will have better neurodevelopmental outcomes. It is also hypothesized that neurobehavioral abnormalities identified at two weeks of age will correlate with neurodevelopmental impairment at 18 months.

3: SPECIFIC Aim III: To determine if common genetic variations in the genes involving narcotic action contribute to the severity of NAS. A DNA sample will be obtained from all infants and analyzed for differences in 3 key genes. This will then be correlated with short-term and long-term outcomes.

DETAILED DESCRIPTION:
1: SPECIFIC Aim I: To compare the short term efficacy of morphine and methadone for the treatment of NAS. One hundred eighty four term infants with a diagnosis of NAS requiring pharmacotherapy will be studied. Infants born to mothers receiving adequate prenatal care and maintained on opioid agonist medication during pregnancy will be eligible. Infants will be randomized to receive either neonatal morphine solution or methadone in a double blind, double dummy design. It is hypothesized that morphine treated infants will require significantly fewer days in the hospital compared to methadone treated infants. While the primary outcome is the total length of initial hospital stay (LOS), total LOS related to NAS, total duration of medical treatment for NAS, the need for a second drug to control symptoms, and infant growth will also be evaluated as important secondary outcomes by medication group assignment.

2. SPECIFIC Aim II: To evaluate the effects of NAS treatment on long-term neurodevelopmental outcome. Infants in both treatment groups will be evaluated at 18 months of age using the Bayley III Scales of Infant Development. It is hypothesized that morphine treated infants will have better neurodevelopmental outcomes at 18 months compared to methadone treated infants. It is also hypothesized that neurobehavioral abnormalities (from either treatment group) identified at two weeks of age using the Neonatal Intensive Care Unit (NICU) Network Neurobehavioral Scale (NNNS) will correlate with neurodevelopmental impairment detected with the Bayley III. Early identification of infants at highest risk for impaired development will facilitate therapeutic interventions to improve outcome and decrease resource utilization.

3: SPECIFIC Aim III: To determine if single nucleotide polymorphisms (SNPs) in genes controlling opioid pharmacodynamics contribute to the severity of NAS. SNP genotyping from cord blood or buccal swabs will be obtained from all infants and correlated with short term outcomes (Aim 1) and neurodevelopment assessments (Aim 2) to confirm that genetic variation plays a major role in the severity and outcome of infants with NAS.

ELIGIBILITY:
Inclusion criteria:

1. Mother receiving methadone or buprenorphine (BPH) from a licensed physician or drug treatment program, or an opioid prescribed by a licensed health care worker for treatment of chronic pain.
2. Need for treatment of NAS by Finnegan Scoring criteria
3. Gestational age >37 weeks at birth defined by best obstetrical estimate
4. Medically stable in the opinion of the Attending Physician
5. Mother receiving "adequate" or "intermediate" prenatal care from a qualified physician or midwife as defined by the Prenatal Care Adequacy Index
6. Singleton pregnancy
7. Mother able to provide informed consent
8. Infant able to take oral medications

Exclusion criteria:

1. Gestation <37 weeks at entry defined by best obstetrical estimate
2. Major congenital abnormalities including genetic syndromes
3. Serious medical illness such as sepsis, asphyxia, seizures, or respiratory failure
4. Mother abusing alcohol during pregnancy (average of 3 or more drinks per week in the last 30 days)
5. Multiple gestations
6. Mother received "inadequate" prenatal care as defined by the Prenatal Care Adequacy Index.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03-05 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Davis, MD, Principal Investigator — Tufts Medical Center; Barry Lester, PhD, Principal Investigator — Women and Infant's Hospital
Locations (8):
- United States (8):
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Women and Infant's Hospital of Rhode Island, Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Wachman EM, Hayes MJ, Brown MS, Paul J, Harvey-Wilkes K, Terrin N, Huggins GS, Aranda JV, Davis JM. Association of OPRM1 and COMT single-nucleotide polymorphisms with hospital length of stay and treatment of neonatal abstinence syndrome. JAMA. 2013 May 1;309(17):1821-7. doi: 10.1001/jama.2013.3411. PMID 23632726
- [Background] Sarkar S, Donn SM. Management of neonatal abstinence syndrome in neonatal intensive care units: a national survey. J Perinatol. 2006 Jan 1;26(1):15-7. doi: 10.1038/sj.jp.7211427. PMID 16355103
- [Background] Lainwala S, Brown ER, Weinschenk NP, Blackwell MT, Hagadorn JI. A retrospective study of length of hospital stay in infants treated for neonatal abstinence syndrome with methadone versus oral morphine preparations. Adv Neonatal Care. 2005 Oct;5(5):265-72. doi: 10.1016/j.adnc.2005.06.003. PMID 16202968
- [Background] Lotsch J, Skarke C, Liefhold J, Geisslinger G. Genetic predictors of the clinical response to opioid analgesics: clinical utility and future perspectives. Clin Pharmacokinet. 2004;43(14):983-1013. doi: 10.2165/00003088-200443140-00003. PMID 15530129
- [Background] Jansson LM, Velez M, Harrow C. The opioid-exposed newborn: assessment and pharmacologic management. J Opioid Manag. 2009 Jan-Feb;5(1):47-55. PMID 19344048
- [Background] Osborn DA, Jeffery HE, Cole MJ. Opiate treatment for opiate withdrawal in newborn infants. Cochrane Database Syst Rev. 2010 Oct 6;(10):CD002059. doi: 10.1002/14651858.CD002059.pub3. PMID 20927730
- [Background] Jones HE, Kaltenbach K, Heil SH, Stine SM, Coyle MG, Arria AM, O'Grady KE, Selby P, Martin PR, Fischer G. Neonatal abstinence syndrome after methadone or buprenorphine exposure. N Engl J Med. 2010 Dec 9;363(24):2320-31. doi: 10.1056/NEJMoa1005359. PMID 21142534
- [Derived] Zankl A, Martin J, Davey JG, Osborn DA. Opioid treatment for opioid withdrawal in newborn infants. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD002059. doi: 10.1002/14651858.CD002059.pub4. PMID 34231914
- [Derived] Czynski AJ, Davis JM, Dansereau LM, Engelhardt B, Marro P, Bogen DL, Hudak ML, Shenberger J, Wachman EM, Oliveira EL, Lester BM. Neurodevelopmental Outcomes of Neonates Randomized to Morphine or Methadone for Treatment of Neonatal Abstinence Syndrome. J Pediatr. 2020 Apr;219:146-151.e1. doi: 10.1016/j.jpeds.2019.12.018. Epub 2020 Jan 24. PMID 31987653
- [Derived] Davis JM, Shenberger J, Terrin N, Breeze JL, Hudak M, Wachman EM, Marro P, Oliveira EL, Harvey-Wilkes K, Czynski A, Engelhardt B, D'Apolito K, Bogen D, Lester B. Comparison of Safety and Efficacy of Methadone vs Morphine for Treatment of Neonatal Abstinence Syndrome: A Randomized Clinical Trial. JAMA Pediatr. 2018 Aug 1;172(8):741-748. doi: 10.1001/jamapediatrics.2018.1307. PMID 29913015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at Tufts Medical Center, Baystate Children's Hospital, Boston Medical Center, Maine Medical Center, Shands Jacksonville Medical Center, University of Pittsburgh Medical Center, Vanderbilt University Medical Center, and Women & Infants Hospital of Rhode Island.
Pre-assignment Details: If infant was diagnosed with NAS (Finnegan score ≥8 on two consecutive occasions, or ≥12 on single assessment) and research pharmacy staff were unavailable for preparation of trial drug, infant could receive one dose of morphine prior to randomization. Dosing was based on weight and Finnegan scores.
Groups:
- Methadone: First line therapy: 0.4mg/mL oral solution, based on weight and symptoms.
  Clinical monitoring: Infants scored using standardized Finnegan system;
  Regimen: Initiated treatment w/ 2 consec. scores ≥8, or 1 score ≥12. Starting doses range 0.3mg/kg/day - 0.9mg/kg/day, divided every 8hrs depending on the severity of Finnegan scores. Doses were increased to max of 0.9mg/kg/day for contd. scores generally >8 caused primarily by worsening NAS, as needed. Weaned by 10% of max dose every 24-48 hours; Medication discontinued once at 25% of max dose.
  Second Line Therapy: Phenobarbital (20mg/kg) was added once infant reached max methadone doses for contd. scores generally >8. Option to re-load w/ 10mg/kg q8-12 hours for 2 more doses if needed for contd. high scores. Maintenance therapy of 5mg/kg/day was initiated 12 - 24hrs after last loading dose. Phenobarbital trough levels monitored, w/ goal levels 20 - 30 mcg/mL. Weaning procedure outlined in protocol.
- Neonatal Morphine Solution: First line therapy: 0.2mg/mL solution, based on weight and symptoms.
  Clinical monitoring: Infants scored using standardized Finnegan system;
  Regimen: Initiated treatment w/ 2 consec. scores ≥8, or 1 score ≥12. Starting doses range 0.3mg/kg/day - 0.9mg/kg/day, divided every 4hrs depending on the severity of Finnegan scores. Doses were increased to max of 0.9mg/kg/day for contd. scores generally >8 caused primarily by worsening NAS, as needed. Weaned by 10% of max dose every 24 - 48 hours; Medication discontinued once at 25% of max dose.
  Second Line Therapy: Phenobarbital (20mg/kg) was added once infant reached max morphine doses for contd. scores generally >8. Option to re-load w/ 10mg/kg q8-12 hours for 2 more doses if needed for contd. high scores. Maintenance therapy of 5mg/kg/day was initiated 12 - 24hrs after last loading dose. Phenobarbital trough levels monitored, w/ goal levels 20 - 30 mcg/mL. Weaning procedure outlined in protocol.
Period: Overall Study
Arm/Group | Methadone | Neonatal Morphine Solution
Started | 59 | 58
Completed | 58 | 58
Not Completed | 1 | 0
Not completed — Parent requested exclusion from analysis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized: Methadone: First line therapy: 0.4mg/mL oral solution, based on weight and symptoms.
  Clinical monitoring: Infants scored using standardized Finnegan system;
  Regimen: Initiated treatment w/ 2 consec. scores ≥8, or 1 score ≥12. Starting doses range 0.3mg/kg/day - 0.9mg/kg/day, divided every 8hrs depending on the severity of Finnegan scores. Doses were increased to max of 0.9mg/kg/day for contd. scores generally >8 caused primarily by worsening NAS, as needed. Weaned by 10% of max dose every 24-48 hours; Medication discontinued once at 25% of max dose.
  Second Line Therapy: Phenobarbital (20mg/kg) was added once infant reached max methadone doses for contd. scores generally >8. Option to re-load w/ 10mg/kg q8-12 hours for 2 more doses if needed for contd. high scores. Maintenance therapy of 5mg/kg/day was initiated 12 - 24hrs after last loading dose. Phenobarbital trough levels monitored, w/ goal levels 20 - 30 mcg/mL. Weaning procedure outlined in protocol.
- Randomized: Neonatal Morphine Solution: First line therapy: 0.2mg/mL solution, based on weight and symptoms.
  Clinical monitoring: Infants scored using standardized Finnegan system;
  Regimen: Initiated treatment w/ 2 consec. scores ≥8, or 1 score ≥12. Starting doses range 0.3mg/kg/day - 0.9mg/kg/day, divided every 4hrs depending on the severity of Finnegan scores. Doses were increased to max of 0.9mg/kg/day for contd. scores generally >8 caused primarily by worsening NAS, as needed. Weaned by 10% of max dose every 24 - 48 hours; Medication discontinued once at 25% of max dose.
  Second Line Therapy: Phenobarbital (20mg/kg) was added once infant reached max morphine doses for contd. scores generally >8. Option to re-load w/ 10mg/kg q8-12 hours for 2 more doses if needed for contd. high scores. Maintenance therapy of 5mg/kg/day was initiated 12 - 24hrs after last loading dose. Phenobarbital trough levels monitored, w/ goal levels 20 - 30 mcg/mL. Weaning procedure outlined in protocol.
- Total: Total of all reporting groups
Arm/Group | Randomized: Methadone | Randomized: Neonatal Morphine Solution | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Customized [Mean (Standard Deviation); unit: days] — Infant mean age upon starting treatment;
  days | 3.2 (1.3) | 3.5 (1.6) | 3.4 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants] — N (%)
  Participants
    Female | 29 | 29 | 58
    Male | 29 | 29 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — N (%)
  Participants
    Infant Race/Ethnicity: White | 46 | 42 | 88
    Infant Race/Ethnicity: Hispanic | 6 | 6 | 12
    Infant Race/Ethnicity: Other | 6 | 10 | 16
Maternal opioid use [Count of Participants; unit: Participants] — N (%)
  Participants
    Buprenorphine | 20 | 19 | 39
    Methadone | 38 | 35 | 73
    Prescription opioids for pain | 0 | 4 | 4
Maternal Smoking Frequency during Pregnancy [Count of Participants; unit: Participants] — N (%)
  Participants
    Smoked >5 cigarettes per day | 33 | 15 | 48
    Unknown/Data Missing | 25 | 43 | 68
Maternal urine toxicology [Count of Participants; unit: Participants] — Positive for at least one illicit substance, N (%)
  Participants
    Positive urine toxicology | 13 | 16 | 29
    Negative urine toxicology | 41 | 33 | 74
    Data Missing | 4 | 9 | 13
Maternal psychiatric diagnoses [Count of Participants; unit: Participants] — N (%)
  Participants
    Psychiatric diagnoses | 42 | 37 | 79
    No psychiatric diagnoses/Unknown | 16 | 21 | 37
Maternal psychiatric medication during pregnancy [Count of Participants; unit: Participants] — N (%)
  Participants
    Psychiatric medication during pregnancy | 20 | 16 | 36
    No psychiatric medication during pregnancy/Unknown | 38 | 42 | 80
Infant mean gestational age [Mean (Standard Deviation); unit: weeks] | 39.2 (1.2) | 39.1 (1.1) | 39.2 (1.2)
Infant birth weight [Mean (Standard Deviation); unit: grams] | 3186 (488) | 3128 (487) | 3146 (486)
Infant APGAR score at 1 minute [Count of Participants; unit: Participants] — Appearance, Pulse, Grimace, Activity, and Respiration (APGAR), a 5-criteria assessment used to summarize the health of the newborn against infant mortality, scored at 1 minute after birth. Each assessment (Appearance, Pulse, Grimace, Activity, Respiration) is scored on a categorical scale of 0, 1 or 2 based on given criteria. All assessment scores are summarized to create the APGAR score (min = 0, max = 10). An APGAR score ≥7 generally indicates a newborn with normal health; An APGAR score ≤3 is generally considered critically low and cause for resuscitation efforts and critical care.
  Participants
    Score ≥7 | 54 | 53 | 107
    Score <7/Data missing | 4 | 5 | 9
Infant mean head circumference [Mean (Standard Deviation); unit: cm] | 33.9 (1.7) | 33.7 (1.8) | 33.8 (1.7)
Infant urine toxicology [Count of Participants; unit: Participants] — N (%)
  Participants
    Positive | 41 | 42 | 83
    Negative | 14 | 14 | 28
    Missing | 3 | 2 | 5
Site of initial care before treatment [Count of Participants; unit: Participants] — by type of care unit
  Participants
    NICU | 3 | 10 | 13
    Newborn Nursery | 55 | 48 | 103
    Other | 0 | 0 | 0
Single dose of morphine prior to randomization [Count of Participants; unit: Participants] — N (%)
  Participants
    Single dose of morphine prior to randomization | 23 | 17 | 40
    No dose of morphine prior to randomization | 35 | 41 | 76
Initial site of NAS care [Count of Participants; unit: Participants] — N (%)
  Participants
    NICU | 17 | 17 | 34
    Special Care Nursery | 9 | 7 | 16
    General Pediatric Unit | 16 | 18 | 34
    Newborn Unit | 16 | 16 | 32
Starting dose of study drug [Count of Participants; unit: Participants] — N (%)
  Participants
    Level I: 0.3 mg/kg/day | 26 | 32 | 58
    Level II: 0.5 mg/kg/day | 25 | 21 | 46
    Level I: 0.7 mg/kg/day | 7 | 5 | 12
Maximum Finnegan score prior to starting treatment [Mean (Standard Deviation); unit: units on a scale] — Finnegan Scoring Tool, a 25-item assessment of infants for Neonatal Abstinence Syndrome (NAS), is used within 24 hrs after birth and subsequently every 4 hours. Each item is scored on varying categorical subscales, scored depending on severity of each sign/symptom (ex. Generalized seizure Yes=8 No=0; Poor feeding Yes=2 No=0). Individually scored items are added to create the total Finnegan score. One score ≥12 or two consecutive scores ≥8 affirms the requirement for pharmacological treatment or increasing treatment dosage. A higher Finnegan score indicates greater NAS severity (min 0 max 50)
  units on a scale | 12.9 (2.9) | 12.6 (2.8) | NA (NA) — Baseline assessment for randomized cohorts only.
Primary feeding during hospitalization [Count of Participants; unit: Participants] — N (%)
  Participants
    Formula only | 22 | 32 | 54
    Breast milk (exclusive or with formula supplement) | 36 | 26 | 62
Maternal Smoking Status during Pregnancy [Count of Participants; unit: Participants]
  Smoked during pregnancy | 49 | 44 | 93
  Did not smoke during pregancy/Data missing | 9 | 14 | 23
Infant APGAR Score at 5 minutes [Count of Participants; unit: Participants] — Appearance, Pulse, Grimace, Activity, and Respiration (APGAR), a 5-criteria assessment used to summarize the health of the newborn against infant mortality, scored at 5 minutes after birth. Each assessment (Appearance, Pulse, Grimace, Activity, Respiration) is scored on a categorical scale of 0, 1 or 2 based on given criteria. All assessment scores are summarized to create the APGAR score (min = 0, max = 10). An APGAR score ≥7 generally indicates a newborn with normal health; An APGAR score ≤3 is generally considered critically low and cause for resuscitation efforts and critical care.
  Participants
    Score ≥7 | 57 | 57 | 114
    Score <7/Data missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay (LOS)
Description: Participants were monitored for the duration of their hospitalization, an expected mean of 22 days.
Time Frame: Participants will be monitored during their entire hospitalization, expected mean 22 days.
Population: Includes infants requiring treatment for NAS who were randomized to either methadone or morphine study intervention. Analysis does not include Standard Clinical Care cohort.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 58 | 58
days | 21.8 (15) | 23.2 (8.8)

2. Secondary Outcome: Length of Hospital Stay (LOS) Due to Neonatal Abstinence Syndrome (NAS)
Description: Participants were monitored for the duration of their hospitalization attributable to NAS only.
Time Frame: Participants were monitored for the duration of their hospitalization, expected mean 22 days.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 58 | 58
days | 18.9 (7.9) | 21.1 (6.9)

3. Secondary Outcome: Length of Treatment (LOT)
Description: Total number of days infant treated with replacement opioids while admitted to the hospital.
Time Frame: Participants were monitored for the duration of their hospitalization.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 58 | 58
days | 14.7 (8.0) | 16.6 (6.9)

4. Secondary Outcome: Maximum Daily Dose of Replacement Opioid
Description: Maximum daily dose of neonatal morphine solution or methadone during the hospitalization
Time Frame: Participants were monitored for the duration of their hospitalization.
Population: Data were not collected due to insufficient funding to carry out data collection.
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Finnegan Score (FS)
Description: Mean Finnegan withdrawal score during the duration of hospitalization.
Time Frame: Participants were monitored during their entire hospitalization
Population: Data were not collected due to insufficient funding to carry out data collection.
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Infants Needing a Second NAS Medication
Description: Number of infants treated with a second medication following protocol, phenobarbital. If the Finnegan Score remained elevated (still scored ≥8 two times consecutively, or still scored once ≥12) despite increasing to a predetermined maximal opioid dose (methadone or morphine), phenobarbital was administered (20-mg/kg loading dose followed by 4-5 mg/kg daily).
Time Frame: Participants were monitored for the duration of their hospitalization, an average of 22 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 58 | 58
Participants | 10 | 17

7. Secondary Outcome: Growth Outcome: Weight Change From Birth to 18 Months
Description: Growth outcome weight (lbs) depicted as difference in averaged weights from birth to 18 month follow-up visit. Standard deviations were averaged between birth and 18 mo time points.
Time Frame: Birth to 18 month follow-up visit
Population: Participants who were continuously enrolled and attended the 18 month follow-up visit for developmental and growth measures.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 46 | 36
lbs | 19.1 (2.5) | 18.7 (2.8)

8. Secondary Outcome: Growth Outcome: Head Circumference at 18 Months
Description: Average head circumference growth outcome at 18 month follow-up visit.
Time Frame: 18 month follow-up visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 46 | 36
cm | 47.8 (2.4) | 48.2 (2.3)

9. Secondary Outcome: Maximum Finnegan Score
Description: Maximum Finnegan score during the hospitalization
Time Frame: Participants monitored for the duration of their hospitalization.
Population: Data were not collected due to insufficient funding to carry out data collection.
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Growth Outcome: Length at 18 Months
Description: Average length (cm) at 18 month follow-up visit.
Time Frame: 18 month follow-up visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 46 | 36
cm | 82.1 (4.6) | 81.7 (5.2)

11. Other Pre Specified Outcome: Cognitive, Language, and Motor Development From 18 Month Bayley III Neurodevelopmental Assessment
Description: The Bayley Scales of Infant and Toddler Development (BSID-III) assesses the development of infants and children (1-42 months) through a series of developmental play tasks, identifying children with developmental delay. Raw scores of completed items are summarized within three distinct scale scores (Cognitive Scale, Language Scale, Motor Scale). Scale scores are each converted to composite scores to determine the child's performance compared with scores of age-matched children of typical development (percentile rank). A higher composite score indicates more ideal developmental outcome (range 40-160). At 18 month follow-up visit, participants were assessed using the BSID-III for cognitive, language and motor scale composite score outcomes.
Time Frame: Assessment at 18 month follow-up visit
Population: Includes subjects who were randomized and remained enrolled at 18 month follow-up visit.
Measure: Mean (Standard Deviation); unit: scores on a scale (Composite)
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 46 | 36
scores on a scale (Composite)
  Cognitive Composite | 100.1 (21.6) | 98.1 (17.2)
  Language Composite | 96.0 (17.1) | 94.2 (18.2)
  Motor Composite | 103.6 (17.3) | 99.1 (17.2)

12. Post Hoc Outcome: Number of Infants Needing a Dose Increase
Description: One Finnegan score ≥12, or two consecutive scores ≥8 affirms the requirement for pharmacological treatment or increasing treatment dosage. If the infant continued to have two consecutive Finnegan Scores ≥8 two times consecutively, or one ≥12, the dose was increased to the next level. (Level I: 0.3 mg/kg/day) (Level II: 0.5 mg/kg/day) (Level III: 0.7 mg/kg/day)
  A higher Finnegan score indicates greater severity of NAS (min 0, max 50).
Time Frame: Participants were monitored for the duration of their hospitalization, an average of 22 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone | Neonatal Morphine Solution
Number analyzed (Participants) | 58 | 58
Participants | 22 | 28

ADVERSE EVENTS:
Time Frame: Participants were monitored for the duration of their hospitalization, an average of 22 days.
Description: Adverse Events and Serious Adverse Events were reported according to standard definitions.
Groups:
- Methadone: Methadone oral solution (0.4mg/mL) for first line therapy. Infants were scored using the standardized Finnegan Scoring Tool and were initiated on treatment with 2 consecutive scores ≥8 or 1 score ≥12. Dosing was weight and symptom based. Starting doses range from 0.3mg/kg/day - 0.9mg/kg/day divided every 8 hours, depending on the severity of the Finnegan scores. To maintain blinding, a "double dummy" design was used - each infant received both methadone/placebo study drug at 0.4 mg/mL and a morphine/placebo study drug at 0.2 mg/mL. Doses were increased to a maximum of 0.9mg/kg/day for continued scores generally >8 caused primarily by worsening NAS, as needed. Infants were weaned by 10% of the maximum dose every 24-48 hours and the medication was discontinued once at 25% of the maximum dose.
- Neonatal Morphine Solution: Neonatal morphine solution (0.2mg/mL) for first line therapy. Infants were scored using the standardized Finnegan Scoring Tool and were initiated on treatment with 2 consecutive scores ≥8 or 1 score ≥12. Dosing was weight and symptom based. Starting doses range from 0.3mg/kg/day - 0.9mg/kg/day divided every 4 hrs, depending on the severity of the Finnegan scores. To maintain blinding, a "double dummy" design was used - each infant received both methadone/placebo study drug at 0.4 mg/mL and a morphine/placebo study drug at 0.2 mg/mL. Doses were increased to a maximum of 0.9mg/kg/day for continued scores generally >8 caused primarily by worsening NAS, as needed. Infants were weaned by 10% of the maximum dose every 24-48 hours and the medication was discontinued once at 25% of the maximum dose.
Arm/Group | Methadone | Neonatal Morphine Solution
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 5/58 | 3/58
Other Adverse Events (participants affected / at risk) | 8/58 | 6/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone (N=58) | Neonatal Morphine Solution (N=58)
Hypothermia, apnea and lethargy (General disorders) | 1 (1) | 0 (0)
Medication Administration Error (Surgical and medical procedures) | 4 (6) | 3 (3) — Includes "medication error by Registered Nurse (RN)", "missed dose by RN", "incorrect dose supplied by pharmacy", and "Delayed escalation doses by RN";
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methadone (N=58) | Neonatal Morphine Solution (N=58)
Apnea and shallow breathing episodes (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Excessive sleepiness/somnolence (Investigations) | 4 (4) | 2 (2)
Lethargy (Investigations) | 0 (0) | 1 (1)
Hypothermia (Investigations) | 2 (2) | 0 (0)
Stridor/desaturation/shalllow breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bradychardia (Cardiac disorders) | 3 (3) | 1 (1)
Poor feeding (Investigations) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT01958476/Prot_SAP_000.pdf